CLINICAL TRIAL: NCT02220920
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Canagliflozin (TA-7284) as add-on to Insulin in Subjects With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety Study of Canagliflozin (TA-7284) in Combination With Insulin in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TA-7284-11
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Results first posted 2016-12-15 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Canagliflozin; Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Canagliflozin (TA-7284) ＋insulin (Experimental)
  Interventions: Drug: Canagliflozin (TA-7284); Drug: Insulin
- Placebo＋insulin (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Insulin

INTERVENTIONS:
Drug: Canagliflozin (TA-7284) — The patients will receive Canagliflozin orally for 16 weeks
  Arms: Canagliflozin (TA-7284) ＋insulin
Drug: Placebo — The patients will receive Placebo orally for 16 weeks
  Arms: Placebo＋insulin
Drug: Insulin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Canagliflozin (TA-7284) in combination with Insulin in patients with type 2 Diabetes for 16 weeks administration.

DETAILED DESCRIPTION:
This is a randomized, 2-arm, parallel group, double blind study to evaluate the efficacy and safety of Canagliflozin (TA-7284) in Japanese patients with type 2 diabetes mellitus, who are receiving treatment with insulin therapy on diet and exercise and have inadequate glycemic control. The patients will receive either TA-7284 100mg or Placebo orally for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who has been receiving a stable dose and regimen of insulin over 12 weeks before administration of investigational dug
* Patients who are under dietary management and taking therapeutic exercise for diabetes over 12 weeks before administration of investigational drug
* Patients with HbA1c of ≥7.5% and <10.5%
* Patients who were not administered diabetes therapeutic drugs prohibited for concomitant use within 12 weeks before administration of investigational drug

Exclusion Criteria:

* Patients with type 1 diabetes mellitus, diabetes mellitus resulting from pancreatic disorder, or secondary diabetes mellitus (Cushing's syndrome, acromegaly, etc.)
* Patients with severe diabetic complications (proliferative diabetic retinopathy, stage 4 nephropathy, or serious diabetic neuropathy)
* Patients with hereditary glucose-galactose malabsorption or primary renal glucosuria
* Patients with systolic blood pressure of ≥160 mmHg or diastolic blood pressure of ≥100 mmHg
* Patients with serious renal or hepatic disease
* Patients with eGFR of <45 mL/min/1.73 m2
* Patients who are the excessive alcohol addicts
* Patients who are pregnant, lactating and probably pregnant patients and patients who can not agree to contraception

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation
Locations (7):
- Japan (7):
  - Reserch site, Chugoku
  - Reserch site, Chūbu
  - Reserch site, Hokkaido
  - Reserch site, Kanto
  - Reserch site, Kinki
  - Reserch site, Kyushu
  - Reserch site, Tōhoku

REFERENCES:
- [Result] Inagaki N, Harashima S, Maruyama N, Kawaguchi Y, Goda M, Iijima H. Efficacy and safety of canagliflozin in combination with insulin: a double-blind, randomized, placebo-controlled study in Japanese patients with type 2 diabetes mellitus. Cardiovasc Diabetol. 2016 Jun 18;15:89. doi: 10.1186/s12933-016-0407-4. PMID 27316668

RESULTS

PARTICIPANT FLOW:
Groups:
- Canagliflozin (TA-7284) ＋Insulin: Canagliflozin, once daily for 16 weeks
- Placebo＋Insulin: Placebo, once daily for 16 weeks
Period: Overall Study
Arm/Group | Canagliflozin (TA-7284) ＋Insulin | Placebo＋Insulin
Started | 76 | 70
Completed | 73 | 67
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Conflict with the stopping criteria | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canagliflozin (TA-7284) ＋Insulin | Placebo＋Insulin | Total
Number analyzed (Participants) | 76 | 70 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 48 | 95
  >=65 years | 29 | 22 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 21 | 53
  Male | 44 | 49 | 93

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline
Time Frame: baseline and Week 16
Population: Full analysis set, last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Canagliflozin (TA-7284) ＋Insulin | Placebo＋Insulin
Number analyzed (Participants) | 76 | 70
Percent | -0.97 (0.08) | 0.13 (0.08)
Statistical Analysis 1: Comparison: Canagliflozin (TA-7284) ＋Insulin vs Placebo＋Insulin; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -1.10, 95% CI 2-sided [-1.33 to -0.87], Standard Error of Mean 0.11

2. Secondary Outcome: Change in Fasting Plasma Glucose
Time Frame: baseline and Week 16
Population: Full analysis set, last observation carried forward. There was a lack of measurement of fasting plasma glucose at the end of treatment visit(Week 4) in one participant who was randomized to "Canagliflozin(TA-7284) + Insulin" group.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Canagliflozin (TA-7284) ＋Insulin | Placebo＋Insulin
Number analyzed (Participants) | 75 | 70
mg/dL | -34.1 (4.8) | -1.4 (5.0)
Statistical Analysis 1: Comparison: Canagliflozin (TA-7284) ＋Insulin vs Placebo＋Insulin; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -32.6, 95% CI 2-sided [-46.3 to -18.9], Standard Error of Mean 6.9

3. Secondary Outcome: Percent Change in Body Weight
Time Frame: baseline and Week 16
Population: Full analysis set, last observation carried forward. There was a lack of measurement of body weight at the end of treatment visit(Week 4) in one participant who was randomized to "Canagliflozin(TA-7284) + Insulin" group.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Canagliflozin (TA-7284) ＋Insulin | Placebo＋Insulin
Number analyzed (Participants) | 75 | 70
percent change | -2.13 (0.25) | 0.24 (0.26)
Statistical Analysis 1: Comparison: Canagliflozin (TA-7284) ＋Insulin vs Placebo＋Insulin; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -2.37, 95% CI 2-sided [-3.09 to -1.65], Standard Error of Mean 0.36

4. Secondary Outcome: Change in Blood Pressure
Time Frame: baseline and Week 16
Population: Full analysis set, last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Canagliflozin (TA-7284) ＋Insulin | Placebo＋Insulin
Number analyzed (Participants) | 76 | 70
mmHg
  Systolic blood pressure | -3.58 (1.14) | -0.40 (1.19)
  Diastolic blood pressure | -1.55 (0.71) | -0.31 (0.74)
Statistical Analysis 1: Comparison: Canagliflozin (TA-7284) ＋Insulin vs Placebo＋Insulin; Test type: Superiority or Other; p = 0.058, ANCOVA; Least-Squares Mean Difference = -3.19, 95% CI 2-sided [-6.49 to 0.11], Standard Error of Mean 1.67 — Estimated P-Value, Least-Squares Mean Difference, Standard Error of the mean, 95% CI are presented for the change from Baseline in systolic blood pressure for week 16
Statistical Analysis 2: Comparison: Canagliflozin (TA-7284) ＋Insulin vs Placebo＋Insulin; Test type: Superiority or Other; p = 0.232, ANCOVA; Least-Squares Mean Difference = -1.24, 95% CI 2-sided [-3.27 to 0.80], Standard Error of Mean 1.03 — Estimated P-Value, Least-Squares Mean Difference, Standard Error of the mean, 95% CI are presented for the change from Baseline in diastolic blood pressure for week 16

5. Secondary Outcome: Percentage of Participants With "Adverse Events" and "Hypoglycemia and Blood Glucose Decreased"
Time Frame: Week 16
Population: Safety analysis set. "Safety Population" reflects the "as treated" population, and one "Canagliflozin (TA-7284) + Insulin" participant actually received "Placebo + Insulin".
Measure: Number; unit: percentage of participants
Arm/Group | Canagliflozin (TA-7284) ＋Insulin | Placebo＋Insulin
Number analyzed (Participants) | 75 | 71
percentage of participants
  adverse events | 68.0 | 64.8
  Hypoglycemia and Blood glucose decreased | 40.0 | 29.6

ADVERSE EVENTS:
Description: "Safety Population" reflects the "as treated" population, and one "Canagliflozin(TA-7284) + Insulin" participant actually received "Placebo + Insulin".
Arm/Group | Canagliflozin (TA-7284) ＋Insulin | Placebo＋Insulin
Serious Adverse Events (participants affected / at risk) | 3/75 | 1/71
Other Adverse Events (participants affected / at risk) | 39/75 | 34/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canagliflozin (TA-7284) ＋Insulin (N=75) | Placebo＋Insulin (N=71)
Cataract (Eye disorders) | 1 | 1
Retinal detachment (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Alcoholic liver disease (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canagliflozin (TA-7284) ＋Insulin (N=75) | Placebo＋Insulin (N=71)
Nasopharyngitis (Infections and infestations) | 12 | 13
Hypoglycaemia (Metabolism and nutrition disorders) | 19 | 15
Pollakiuria (Renal and urinary disorders) | 4 | 1
Blood glucose decreased (Investigations) | 20 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other